CLINICAL TRIAL: NCT04866888
Title: Short and Intermediate Term Outcomes of Uterine Conservation After Cesarian Section in Cases of Placenta Accreta Spectrum
Brief Title: Placenta Accreta Spectrum Outcome After Uterine Conservation
Acronym: PAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H.R1987
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Placenta Accreta Spectrum
Keywords: PAS
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Uterus will be incised 5mm above the placenta bulge. Uterine exteriorization followed by pealing of amniotic membranes to reach an accessible pole of the placenta to detect a plan of cleavage behind it. The independent hand of the surgeon passed through the previous plan from points of least resistance to high resistance. The defect will be repaired from the inner aspect of the uterus via running sutures using Vicryl (1-0) on a round needle, 45mm. the suture will pass from one edge to hitch the bed and pass to the other edge till we completely close the defect subsequently, controlling the bleeding. Uterine scar closure by running sutures in two layers, where the first layer compresses the placental bed defect externally. After 3 months ultrasound and out-patient hysteroscopy will be done to check for any uterine abnormalities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pregnant women with placenta accreta spectrum (Experimental): Bladder will be dissected and mobilized down to the vagina after skeletonization and securing of bridging vessels either by electro-coagulation or ligation. Uterus will be incised 5mm above the placenta bulge, delivering the fetus followed by Carbetocin 100 microgram /1 ml intravascular. Repair of the uterine wall defect will be done. If extrauterine bleeding is excessive we may revert to internal iliac artery ligation followed by insertion of intra-peritoneal drain and regular abdominal wall closure.
  After 3 months from delivery, ultrasound with different modalities will be done to all patients and outpatient hysteroscopy if symptomatic patients or with abnormal sonography.
  Interventions: Procedure: closure of the uterine wall defect; Diagnostic Test: ultrasound; Diagnostic Test: outpatient hysteroscopy

INTERVENTIONS:
Procedure: closure of the uterine wall defect — Uterine exteriorization followed by pealing of amniotic membranes to reach an accessible pole of the placenta to detect a plan of cleavage behind it. The independent hand of the surgeon passed through the previous plan from points of least resistance to high resistance. The defect will be repaired from the inner aspect of the uterus via running sutures using Vicryl (1-0) on a round needle, 45mm. the suture will pass from one edge to hitch the bed and pass to the other edge till we completely close the defect subsequently, controlling the bleeding. Uterine scar closure by running sutures in two layers, where the first layer compresses the placental bed defect externally.
  Other Names: double compression sutures
Diagnostic Test: ultrasound — Before the procedure transabdominal and transvaginal ultrasound will be done to diagnose PAS and to map the uterine wall defects.
  After 3 months,Transabdominal and transvaginal ultrasound with different modalities to assess the uterine wall, the cavity, endometrium, myometrium and the cervix. Isthmocele will be defined as a defect at uterine wall where residual myometrium thickness and ratio between residual myometrium and total myometrium thickness will be measured and recorded. The shape of the isthmocele will be also recorded.
Diagnostic Test: outpatient hysteroscopy — Office hysteroscope will be done after patient consent to evaluate the uterine cavity if the patient is symptomatic or with abnormal sonography. It will be performed in the proliferative phase of the menstrual cycle. Non-steroidal anti-inflammatory will be given one hour before the procedure, then the patient will be in lithotomy position. Following aseptic rules, the rigid 4 mm hysteroscope will be inserted into the uterus through the cervix without using speculum nor tenaculum. Any pathology will be identified, and data will be recorded.
  Other Names: office hysteroscopy

SUMMARY:
study will be carried out on patients with placenta accreta spectrum having done uterine conservation and recording immediate outcome of conservation regarding success of the procedure, amount of blood loss and amount of blood transfused and followed up to check the return of menses, any uterine abnormalities by ultrasound or hysteroscopy especially isthmocele and intrauterine synechia.

DETAILED DESCRIPTION:
After institutional review board approval and written informed consent, recruited cases will be subjected to the following:

1. Data registration including:

   * Age.
   * Obstetric history including gravidity, parity, number of previous cesarean deliveries, and number and gender of living children.
   * Details of the current pregnancy including duration in menstrual weeks, any problems encountered during its course.
   * Desire for future fertility.
   * Medical, surgical, and medication history.
2. Anthropometry including weight, height, and body mass index (BMI) before pregnancy and at the time of operation.
3. General examination including vital signs, and signs of any associated problems.
4. Routine laboratory investigations with particular emphasis on complete blood count, Coagulation profile and including blood glucose level, renal and liver function tests.
5. Detailed sonographic examination to evaluate fetal biometry, and wellbeing rule out exclusion factors, and confirm diagnosis of PAS and assess the degree of invasion, and its severity using both trans-abdominal transducer with frequency of 2-5 megahertz (MHZ) and trans-vaginal transducer with frequency of 4-10 MHZ.

Intraoperative details will be documented. Follow up of patients will be recorded. Sample size was calculated by estimating a single proportion distribution at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed sonographically to have placenta accreta spectrum.

  * Pregnancy is singleton and fetus is alive.
  * Elective caesarean section done from 35 gestational weeks.

Exclusion Criteria:

* • Patients requesting hysterectomy.

  * Coexisting uterine pathology such as fibroids or gynaecological malignancies.
  * Patients with bleeding diathesis.
  * Morbid obesity of BMI >40.
  * Patients having labour pains or vaginal bleeding before scheduled intervention.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant female patient
Enrollment: 120 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
date of resumed menses | from 2 weeks to 6 months after surgery
  calculate the duration from surgery until menses returns
menstrual abnormalities | from 2 to 6 months after surgery
  record type of menstrual abnormalities if present such as amenorrhea, oligomenorrhea and dysmenorrhea
abnormal uterine bleeding | from 2 to 6 months after surgery
  record the presence of abnormal uterine bleeding after the return of menses such as intermenstrual bleeding, menorrhagia
pelvic pain | from 2 to 6 months after surgery
  record the presence of pelvic pain and its duration
isthmocele | from 3 to 6 months after surgery
  trans-vaginal and trans-abdominal ultrasound will be done to record the presence of isthmocele, its shape and ratio between residual myometrium and total myometrium
intrauterine adhesions | from 3 to 6 months after surgery
  outpatient hysteroscopy will be done to symptomatic patients after consent in order to check uterine cavity recording the presence of intrauterine adhesions, and categorization of adhesions according to american fertility society into mild, moderate and severe
puerperal blood loss | 48 hours until 2 months after surgery
  recording the duration of blood loss during puerperium and average number of tampons changed per day
contraception use | intraoperative until 5 months after surgery
  recording method of contraception used
fibrosis | from 3 to 6 months after surgery
  grey scale ultrasound will be done to record size of intra-myometrium fibrosis

SECONDARY OUTCOMES:
operation time | intraoperative
  recording total time of the surgery
repair time | intraoperative
  recording length of defect repair from placental separation until uterine wall closure
Estimated blood loss | intraoperative
  recording amount of blood loss
packed red blood cells transfusion | intraoperative until 24 hours after surgery
  recording amount of red blood cell transfused
fresh frozen plasma (FFP) transfusion | intraoperative until 24 hours postoperative
  recording amount of FFP transfusion
bladder injury | intraoperative until 2 weeks post operative
  recording if there was an injury to the bladder
ureter injury | intraoperative until 2 weeks post operative
  recording if there was an injury to the ureter
bowel injury | intraoperative until 2 weeks post operative
  recording if there was an injury to the bowel
surgical site infection | 24 hours until 1 month after surgery
  record the presence of wound infection
urine output | intraoperative
  recording amount of urine output
internal iliac artery ligation | intraoperative
  recording if the internal iliac artery ligated whether it was unilateral or bilateral
pre-operative hemoglobin | preoperative
  recording amount of hemoglobin
post-operative hemoglobin | postoperative within 6 hours from surgery
  recording amount of hemoglobin
hospital stay | postoperative until 10 days after surgery
  recording duration of hospital stay after surgery
ICU admission | immediate postoperative until 5 days after surgery
  recording the number of patients admitted to the ICU
intermediate care admission | recording the number of patients admitted to the ICU
  recording the number of patients admitted to the intermediate care
surgical diagnosis | intraoperative
  document the type of placenta accreta spectrum whether it is accreta, increta or percreta and area of the uterus where the placental invade

CONTACTS AND LOCATIONS:
Overall Officials: Mervat S Al-sedik, MD, Study Chair — faculty of medicine department of obstetrics and gyneacology
Locations (1):
- Faculty of Medicine, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual patient data (IPD) that underlies results in publication
Supporting Information: Study Protocol, SAP
Time Frame: after publication for 1 month
Access Criteria: it will be shared with obstetricians and gynecologists

REFERENCES:
- [Derived] Elshorbagy OY, Hamdy MA. Conservative surgical repair of placenta increta invading into uterine septum: case report. J Med Case Rep. 2024 Nov 18;18(1):549. doi: 10.1186/s13256-024-04814-7. PMID 39551821